CLINICAL TRIAL: NCT02338232
Title: Pilot Study of Telmisartan (Micardis) For the Prevention of Acute Graft vs. Host Disease Post Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Study of TelmisartanFor the Prevention of Acute GVHD Post Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro5465
Record Dates: First submitted 2015-01-05; First posted 2015-01-14 (Estimated); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: GVHD
MeSH Terms: interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 160 mg Telmisartan (Experimental): 60 patients will receive 160 of Telmisartan (2 80 mg tablets) for 101 days
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis

SUMMARY:
This is single-center, open-label, prospective study of telmisartan for the prevention of acute GVHD in approximately 60 subjects undergoing allogeneic HCT for treatment of a hematologic malignancy.

DETAILED DESCRIPTION:
This is single-center, open-label, prospective study of telmisartan for the prevention of acute GVHD in approximately 60 subjects undergoing allogeneic HCT for treatment of a hematologic malignancy. Subjects will receive 160 mg Micardis brand telmisartan once daily, starting 2 days prior to HCT (day -2). Once the patient is discharged post-HCT, treatment will continue through Day +98 post-HCT for a total of 101 days. After treatment discontinuation on or before day +98 post-HCT, subjects will be followed for up to 6 months for primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of:

  * Acute myeloid or lymphoid leukemia in remission,
  * Myelodysplastic syndrome,
  * Chronic lymphoid leukemia,
  * Non-Hodgkin lymphoma,
  * Hodgkin lymphoma,
  * Chronic myeloid leukemia in chronic or accelerated phase,
  * Myeloproliferative disorder, or
  * Multiple myeloma
* Undergoing allogeneic HSC transplantation from a related or unrelated donor matched at least at 7 of 8 of the HLA-A, -B, -C, and DR loci ("8/8" or "7/8" match)
* Undergoing allogeneic HSC transplantation after a myeloablative TBI-, busulfan-, or (non-myeloablative) melphalan-based pre-transplant conditioning regimen. Regimens for transplantation will include at one of the following agents, given in conjunction with fludarabine or cyclophosphamide:

  * Busulfan 130 mg/m2 iv daily x 2 (reduced intensity) or 4 days
  * TBI 150 cGy bid x8 doses (1200 Gy)
  * Melphalan 140 mg/m2. (Although melphalan is not a myeloablative regimen, it results in clinically significant mucositis and patients receiving this medication will be of considerable interest in the analysis of these data.)
* Male or female patient age 18 years or older
* Karnofsky performance status > 70% at time of initiation of pre-transplant conditioning
* Transplantation-specific co-morbidity score of <5 at time of initiation of pre-transplant conditioning
* Patients taking antihypertensive medications (including telmisartan) are eligible but the patient must discontinue treatment at least 48 hours prior to first dose of study medication
* Capable of giving informed consent and having signed the informed consent form

Exclusion Criteria:

* Inability to provide informed consent
* Subjects with known heart failure, advanced renal impairment requiring renal replacement therapy, or liver failure although these patients would most likely not be eligible for HCT.
* Subjects taking ACE inhibitors, potassium supplements, or spironolactone (or any other potassium-sparing diuretics) who cannot discontinue use prior to initiation of study treatment OR who require a high-potassium diet
* Patient unable to discontinue current hypertension medication for medical or other reasons for two days prior to starting telmisartan
* Chronic symptomatic hypotension, volume depletion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rowley, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Hill GR, Ferrara JL. The primacy of the gastrointestinal tract as a target organ of acute graft-versus-host disease: rationale for the use of cytokine shields in allogeneic bone marrow transplantation. Blood. 2000 May 1;95(9):2754-9. PMID 10779417
- [Background] Chen X, Dodge J, Komorowski R, Drobyski WR. A critical role for the retinoic acid signaling pathway in the pathophysiology of gastrointestinal graft-versus-host disease. Blood. 2013 May 9;121(19):3970-80. doi: 10.1182/blood-2012-08-445130. Epub 2013 Mar 25. PMID 23529927
- [Background] Eriguchi Y, Takashima S, Oka H, Shimoji S, Nakamura K, Uryu H, Shimoda S, Iwasaki H, Shimono N, Ayabe T, Akashi K, Teshima T. Graft-versus-host disease disrupts intestinal microbial ecology by inhibiting Paneth cell production of alpha-defensins. Blood. 2012 Jul 5;120(1):223-31. doi: 10.1182/blood-2011-12-401166. Epub 2012 Apr 24. PMID 22535662
- [Background] Blazar BR, Murphy WJ, Abedi M. Advances in graft-versus-host disease biology and therapy. Nat Rev Immunol. 2012 May 11;12(6):443-58. doi: 10.1038/nri3212. PMID 22576252
- [Background] Wolf D, von Lilienfeld-Toal M, Wolf AM, Schleuning M, von Bergwelt-Baildon M, Held SA, Brossart P. Novel treatment concepts for graft-versus-host disease. Blood. 2012 Jan 5;119(1):16-25. doi: 10.1182/blood-2011-08-339465. Epub 2011 Sep 26. PMID 21948301
- [Background] Choi S, Reddy P. Graft-versus-host disease. Panminerva Med. 2010 Jun;52(2):111-24. PMID 20517195
- [Background] Ringden O, Shrestha S, da Silva GT, Zhang MJ, Dispenzieri A, Remberger M, Kamble R, Freytes CO, Gale RP, Gibson J, Gupta V, Holmberg L, Lazarus H, McCarthy P, Meehan K, Schouten H, Milone GA, Lonial S, Hari PN. Effect of acute and chronic GVHD on relapse and survival after reduced-intensity conditioning allogeneic transplantation for myeloma. Bone Marrow Transplant. 2012 Jun;47(6):831-7. doi: 10.1038/bmt.2011.192. Epub 2011 Sep 26. PMID 21946381
- [Background] Lee SJ, Klein JP, Barrett AJ, Ringden O, Antin JH, Cahn JY, Carabasi MH, Gale RP, Giralt S, Hale GA, Ilhan O, McCarthy PL, Socie G, Verdonck LF, Weisdorf DJ, Horowitz MM. Severity of chronic graft-versus-host disease: association with treatment-related mortality and relapse. Blood. 2002 Jul 15;100(2):406-14. doi: 10.1182/blood.v100.2.406. PMID 12091329
- [Background] Signori A, Crocchiolo R, Oneto R, Sacchi N, Sormani MP, Fagioli F, Rambaldi A, Ciceri F, Bacigalupo A. Chronic GVHD is associated with lower relapse risk irrespective of stem cell source among patients receiving transplantation from unrelated donors. Bone Marrow Transplant. 2012 Nov;47(11):1474-8. doi: 10.1038/bmt.2012.58. Epub 2012 Apr 2. PMID 22465976
- [Background] Patterson AE, Korngold R. Infusion of select leukemia-reactive TCR Vbeta+ T cells provides graft-versus-leukemia responses with minimization of graft-versus-host disease following murine hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2001;7(4):187-96. doi: 10.1053/bbmt.2001.v7.pm11349805.
- [Background] Fanning SL, Zilberberg J, Stein J, Vazzana K, Berger SA, Korngold R, Friedman TM. Unraveling graft-versus-host disease and graft-versus-leukemia responses using TCR Vbeta spectratype analysis in a murine bone marrow transplantation model. J Immunol. 2013 Jan 1;190(1):447-57. doi: 10.4049/jimmunol.1201641. Epub 2012 Nov 30. PMID 23203931
- [Background] Komanduri KV. Targeting neovascularization in GVHD. Blood. 2013 Apr 25;121(17):3303-4. doi: 10.1182/blood-2013-01-480483. PMID 23620570
- [Background] Leonhardt F, Grundmann S, Behe M, Bluhm F, Dumont RA, Braun F, Fani M, Riesner K, Prinz G, Hechinger AK, Gerlach UV, Dierbach H, Penack O, Schmitt-Graff A, Finke J, Weber WA, Zeiser R. Inflammatory neovascularization during graft-versus-host disease is regulated by alphav integrin and miR-100. Blood. 2013 Apr 25;121(17):3307-18. doi: 10.1182/blood-2012-07-442665. Epub 2013 Jan 17. PMID 23327924
- [Background] Penack O, Socie G, van den Brink MR. The importance of neovascularization and its inhibition for allogeneic hematopoietic stem cell transplantation. Blood. 2011 Apr 21;117(16):4181-9. doi: 10.1182/blood-2010-10-312934. Epub 2011 Jan 21. PMID 21258010
- [Background] Penack O, Henke E, Suh D, King CG, Smith OM, Na IK, Holland AM, Ghosh A, Lu SX, Jenq RR, Liu C, Murphy GF, Lu TT, May C, Scheinberg DA, Gao DC, Mittal V, Heller G, Benezra R, van den Brink MR. Inhibition of neovascularization to simultaneously ameliorate graft-vs-host disease and decrease tumor growth. J Natl Cancer Inst. 2010 Jun 16;102(12):894-908. doi: 10.1093/jnci/djq172. Epub 2010 May 12. PMID 20463307
- [Background] Petrovic A, Alpdogan O, Willis LM, Eng JM, Greenberg AS, Kappel BJ, Liu C, Murphy GJ, Heller G, van den Brink MR. LPAM (alpha 4 beta 7 integrin) is an important homing integrin on alloreactive T cells in the development of intestinal graft-versus-host disease. Blood. 2004 Feb 15;103(4):1542-7. doi: 10.1182/blood-2003-03-0957. Epub 2003 Oct 16. PMID 14563643
- [Background] Reshef R, Luger SM, Hexner EO, Loren AW, Frey NV, Nasta SD, Goldstein SC, Stadtmauer EA, Smith J, Bailey S, Mick R, Heitjan DF, Emerson SG, Hoxie JA, Vonderheide RH, Porter DL. Blockade of lymphocyte chemotaxis in visceral graft-versus-host disease. N Engl J Med. 2012 Jul 12;367(2):135-45. doi: 10.1056/NEJMoa1201248. PMID 22784116
- [Background] Engelhardt BG, Jagasia M, Savani BN, Bratcher NL, Greer JP, Jiang A, Kassim AA, Lu P, Schuening F, Yoder SM, Rock MT, Crowe JE Jr. Regulatory T cell expression of CLA or alpha(4)beta(7) and skin or gut acute GVHD outcomes. Bone Marrow Transplant. 2011 Mar;46(3):436-42. doi: 10.1038/bmt.2010.127. Epub 2010 May 31. PMID 20577222
- [Background] Engelhardt BG, Sengsayadeth SM, Jagasia M, Savani BN, Kassim AA, Lu P, Shyr Y, Yoder SM, Rock MT, Crowe JE Jr. Tissue-specific regulatory T cells: biomarker for acute graft-vs-host disease and survival. Exp Hematol. 2012 Dec;40(12):974-982.e1. doi: 10.1016/j.exphem.2012.08.002. Epub 2012 Aug 10. PMID 22885125
- [Background] Brunstein CG, Miller JS, Cao Q, McKenna DH, Hippen KL, Curtsinger J, Defor T, Levine BL, June CH, Rubinstein P, McGlave PB, Blazar BR, Wagner JE. Infusion of ex vivo expanded T regulatory cells in adults transplanted with umbilical cord blood: safety profile and detection kinetics. Blood. 2011 Jan 20;117(3):1061-70. doi: 10.1182/blood-2010-07-293795. Epub 2010 Oct 15. PMID 20952687
- [Background] Liu Z, Zhao Y, Wei F, Ye L, Lu F, Zhang H, Diao Y, Song H, Qi Z. Treatment with telmisartan/rosuvastatin combination has a beneficial synergistic effect on ameliorating Th17/Treg functional imbalance in hypertensive patients with carotid atherosclerosis. Atherosclerosis. 2014 Mar;233(1):291-9. doi: 10.1016/j.atherosclerosis.2013.12.004. Epub 2014 Jan 10. PMID 24495792
- [Background] Mihaescu A, Santen S, Jeppsson B, Thorlacius H. Rho kinase signalling mediates radiation-induced inflammation and intestinal barrier dysfunction. Br J Surg. 2011 Jan;98(1):124-31. doi: 10.1002/bjs.7279. Epub 2010 Sep 29. PMID 20882561
- [Background] Arab HH, Al-Shorbagy MY, Abdallah DM, Nassar NN. Telmisartan attenuates colon inflammation, oxidative perturbations and apoptosis in a rat model of experimental inflammatory bowel disease. PLoS One. 2014 May 15;9(5):e97193. doi: 10.1371/journal.pone.0097193. eCollection 2014. PMID 24831514
- [Background] Kobayashi N, Ohno T, Yoshida K, Fukushima H, Mamada Y, Nomura M, Hirata H, Machida Y, Shinoda M, Suzuki N, Matsuoka H. Cardioprotective mechanism of telmisartan via PPAR-gamma-eNOS pathway in dahl salt-sensitive hypertensive rats. Am J Hypertens. 2008 May;21(5):576-81. doi: 10.1038/ajh.2008.27. Epub 2008 Mar 20. PMID 18437150
- [Background] Iyengar S, Zhan C, Lu J, Korngold R, Schwartz DH. Treatment with a rho kinase inhibitor improves survival from graft-versus-host disease in mice after MHC-haploidentical hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2014 Aug;20(8):1104-11. doi: 10.1016/j.bbmt.2014.04.029. Epub 2014 May 2. PMID 24796280
- [Background] Song EK, Yim JM, Yim JY, Song MY, Rho HW, Yim SK, Jeon SY, Kim HS, Yhim HY, Lee NR, Kwak JY, Sohn MH, Park HS, Jang KY, Yim CY. Rosiglitazone prevents graft-versus-host disease (GVHD). Transpl Immunol. 2012 Oct;27(2-3):128-37. doi: 10.1016/j.trim.2012.09.001. Epub 2012 Sep 13. PMID 22982856
- [Background] Walcher D, Hess K, Heinz P, Petscher K, Vasic D, Kintscher U, Clemenz M, Hartge M, Raps K, Hombach V, Marx N. Telmisartan inhibits CD4-positive lymphocyte migration independent of the angiotensin type 1 receptor via peroxisome proliferator-activated receptor-gamma. Hypertension. 2008 Feb;51(2):259-66. doi: 10.1161/HYPERTENSIONAHA.107.099028. Epub 2007 Dec 24. PMID 18158351
- [Background] Cianchetti S, Del Fiorentino A, Colognato R, Di Stefano R, Franzoni F, Pedrinelli R. Anti-inflammatory and anti-oxidant properties of telmisartan in cultured human umbilical vein endothelial cells. Atherosclerosis. 2008 May;198(1):22-8. doi: 10.1016/j.atherosclerosis.2007.09.013. Epub 2007 Oct 22. PMID 17950296
- [Background] Siragusa M, Sessa WC. Telmisartan exerts pleiotropic effects in endothelial cells and promotes endothelial cell quiescence and survival. Arterioscler Thromb Vasc Biol. 2013 Aug;33(8):1852-60. doi: 10.1161/ATVBAHA.112.300985. Epub 2013 May 23. PMID 23702662
- [Background] Usui T, Sugisaki K, Iriyama A, Yokoo S, Yamagami S, Nagai N, Ishida S, Amano S. Inhibition of corneal neovascularization by blocking the angiotensin II type 1 receptor. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4370-6. doi: 10.1167/iovs.07-0964. PMID 18829859
- [Background] Nagai N, Noda K, Urano T, Kubota Y, Shinoda H, Koto T, Shinoda K, Inoue M, Shiomi T, Ikeda E, Tsubota K, Suda T, Oike Y, Ishida S. Selective suppression of pathologic, but not physiologic, retinal neovascularization by blocking the angiotensin II type 1 receptor. Invest Ophthalmol Vis Sci. 2005 Mar;46(3):1078-84. doi: 10.1167/iovs.04-1101. PMID 15728568
- [Background] Riento K, Ridley AJ. Rocks: multifunctional kinases in cell behaviour. Nat Rev Mol Cell Biol. 2003 Jun;4(6):446-56. doi: 10.1038/nrm1128. PMID 12778124
- [Background] Yoneda A, Multhaupt HA, Couchman JR. The Rho kinases I and II regulate different aspects of myosin II activity. J Cell Biol. 2005 Aug 1;170(3):443-53. doi: 10.1083/jcb.200412043. Epub 2005 Jul 25. PMID 16043513
- [Background] Wang Y, Zheng XR, Riddick N, Bryden M, Baur W, Zhang X, Surks HK. ROCK isoform regulation of myosin phosphatase and contractility in vascular smooth muscle cells. Circ Res. 2009 Feb 27;104(4):531-40. doi: 10.1161/CIRCRESAHA.108.188524. Epub 2009 Jan 8. PMID 19131646
- [Background] Vicari RM, Chaitman B, Keefe D, Smith WB, Chrysant SG, Tonkon MJ, Bittar N, Weiss RJ, Morales-Ballejo H, Thadani U; Fasudil Study Group. Efficacy and safety of fasudil in patients with stable angina: a double-blind, placebo-controlled, phase 2 trial. J Am Coll Cardiol. 2005 Nov 15;46(10):1803-11. doi: 10.1016/j.jacc.2005.07.047. Epub 2005 Oct 19. PMID 16286163
- [Background] Shimokawa H, Hiramori K, Iinuma H, Hosoda S, Kishida H, Osada H, Katagiri T, Yamauchi K, Yui Y, Minamino T, Nakashima M, Kato K. Anti-anginal effect of fasudil, a Rho-kinase inhibitor, in patients with stable effort angina: a multicenter study. J Cardiovasc Pharmacol. 2002 Nov;40(5):751-61. doi: 10.1097/00005344-200211000-00013. PMID 12409984
- [Background] Fukumoto Y, Mohri M, Inokuchi K, Ito A, Hirakawa Y, Masumoto A, Hirooka Y, Takeshita A, Shimokawa H. Anti-ischemic effects of fasudil, a specific Rho-kinase inhibitor, in patients with stable effort angina. J Cardiovasc Pharmacol. 2007 Mar;49(3):117-21. doi: 10.1097/FJC.0b013e31802ef532. PMID 17414222
- [Background] Otsuka T, Ibuki C, Suzuki T, Ishii K, Kodani E, Atarashi H, Kishida H, Takano T. Vasodilatory effect of subsequent administration of fasudil, a rho-kinase inhibitor, surpasses that of nitroglycerin at the concentric coronary stenosis in patients with stable angina pectoris. Circ J. 2006 Apr;70(4):402-8. doi: 10.1253/circj.70.402. PMID 16565555
- [Background] Masumoto A, Mohri M, Shimokawa H, Urakami L, Usui M, Takeshita A. Suppression of coronary artery spasm by the Rho-kinase inhibitor fasudil in patients with vasospastic angina. Circulation. 2002 Apr 2;105(13):1545-7. doi: 10.1161/hc1002.105938. PMID 11927519
- [Background] Mohri M, Shimokawa H, Hirakawa Y, Masumoto A, Takeshita A. Rho-kinase inhibition with intracoronary fasudil prevents myocardial ischemia in patients with coronary microvascular spasm. J Am Coll Cardiol. 2003 Jan 1;41(1):15-9. doi: 10.1016/s0735-1097(02)02632-3. PMID 12570938
- [Background] Inokuchi K, Ito A, Fukumoto Y, Matoba T, Shiose A, Nishida T, Masuda M, Morita S, Shimokawa H. Usefulness of fasudil, a Rho-kinase inhibitor, to treat intractable severe coronary spasm after coronary artery bypass surgery. J Cardiovasc Pharmacol. 2004 Sep;44(3):275-7. doi: 10.1097/01.fjc.0000134775.76636.3f. PMID 15475822
- [Background] Kishi T, Hirooka Y, Masumoto A, Ito K, Kimura Y, Inokuchi K, Tagawa T, Shimokawa H, Takeshita A, Sunagawa K. Rho-kinase inhibitor improves increased vascular resistance and impaired vasodilation of the forearm in patients with heart failure. Circulation. 2005 May 31;111(21):2741-7. doi: 10.1161/CIRCULATIONAHA.104.510248. PMID 15927989
- [Background] Witzenrath M, Ahrens B, Schmeck B, Kube SM, Hippenstiel S, Rosseau S, Hamelmann E, Suttorp N, Schutte H. Rho-kinase and contractile apparatus proteins in murine airway hyperresponsiveness. Exp Toxicol Pathol. 2008 Jun;60(1):9-15. doi: 10.1016/j.etp.2008.03.002. Epub 2008 Apr 22. PMID 18434112
- [Background] Noma K, Rikitake Y, Oyama N, Yan G, Alcaide P, Liu PY, Wang H, Ahl D, Sawada N, Okamoto R, Hiroi Y, Shimizu K, Luscinskas FW, Sun J, Liao JK. ROCK1 mediates leukocyte recruitment and neointima formation following vascular injury. J Clin Invest. 2008 May;118(5):1632-44. doi: 10.1172/JCI29226. PMID 18414683
- [Background] Lammermann T, Bader BL, Monkley SJ, Worbs T, Wedlich-Soldner R, Hirsch K, Keller M, Forster R, Critchley DR, Fassler R, Sixt M. Rapid leukocyte migration by integrin-independent flowing and squeezing. Nature. 2008 May 1;453(7191):51-5. doi: 10.1038/nature06887. PMID 18451854
- [Background] Smith A, Bracke M, Leitinger B, Porter JC, Hogg N. LFA-1-induced T cell migration on ICAM-1 involves regulation of MLCK-mediated attachment and ROCK-dependent detachment. J Cell Sci. 2003 Aug 1;116(Pt 15):3123-33. doi: 10.1242/jcs.00606. Epub 2003 Jun 10. PMID 12799414
- [Background] van Buul JD, Hordijk PL. Signaling in leukocyte transendothelial migration. Arterioscler Thromb Vasc Biol. 2004 May;24(5):824-33. doi: 10.1161/01.ATV.0000122854.76267.5c. Epub 2004 Feb 19. PMID 14976004
- [Background] Benais-Pont G, Punn A, Flores-Maldonado C, Eckert J, Raposo G, Fleming TP, Cereijido M, Balda MS, Matter K. Identification of a tight junction-associated guanine nucleotide exchange factor that activates Rho and regulates paracellular permeability. J Cell Biol. 2003 Mar 3;160(5):729-40. doi: 10.1083/jcb.200211047. Epub 2003 Feb 25. PMID 12604587
- [Background] Li B, Zhao WD, Tan ZM, Fang WG, Zhu L, Chen YH. Involvement of Rho/ROCK signalling in small cell lung cancer migration through human brain microvascular endothelial cells. FEBS Lett. 2006 Jul 24;580(17):4252-60. doi: 10.1016/j.febslet.2006.06.056. Epub 2006 Jun 30. PMID 16828752
- [Background] Nohria A, Grunert ME, Rikitake Y, Noma K, Prsic A, Ganz P, Liao JK, Creager MA. Rho kinase inhibition improves endothelial function in human subjects with coronary artery disease. Circ Res. 2006 Dec 8;99(12):1426-32. doi: 10.1161/01.RES.0000251668.39526.c7. Epub 2006 Nov 9. PMID 17095725
- [Background] Bardi G, Niggli V, Loetscher P. Rho kinase is required for CCR7-mediated polarization and chemotaxis of T lymphocytes. FEBS Lett. 2003 May 8;542(1-3):79-83. doi: 10.1016/s0014-5793(03)00351-x. PMID 12729902
- [Background] Lee JH, Katakai T, Hara T, Gonda H, Sugai M, Shimizu A. Roles of p-ERM and Rho-ROCK signaling in lymphocyte polarity and uropod formation. J Cell Biol. 2004 Oct 25;167(2):327-37. doi: 10.1083/jcb.200403091. PMID 15504914
- [Background] Xue F, Takahara T, Yata Y, Xia Q, Nonome K, Shinno E, Kanayama M, Takahara S, Sugiyama T. Blockade of Rho/Rho-associated coiled coil-forming kinase signaling can prevent progression of hepatocellular carcinoma in matrix metalloproteinase-dependent manner. Hepatol Res. 2008 Aug;38(8):810-7. doi: 10.1111/j.1872-034X.2008.00333.x. Epub 2008 May 27. PMID 18507693
- [Background] Wong CC, Wong CM, Ko FC, Chan LK, Ching YP, Yam JW, Ng IO. Deleted in liver cancer 1 (DLC1) negatively regulates Rho/ROCK/MLC pathway in hepatocellular carcinoma. PLoS One. 2008 Jul 23;3(7):e2779. doi: 10.1371/journal.pone.0002779. PMID 18648664
- [Background] Ogawa T, Tashiro H, Miyata Y, Ushitora Y, Fudaba Y, Kobayashi T, Arihiro K, Okajima M, Asahara T. Rho-associated kinase inhibitor reduces tumor recurrence after liver transplantation in a rat hepatoma model. Am J Transplant. 2007 Feb;7(2):347-55. doi: 10.1111/j.1600-6143.2006.01647.x. Epub 2007 Jan 4. PMID 17229077
- [Background] Wang DS, Dou KF, Li KZ, Song ZS. Enhancement of migration and invasion of hepatoma cells via a Rho GTPase signaling pathway. World J Gastroenterol. 2004 Jan 15;10(2):299-302. doi: 10.3748/wjg.v10.i2.299. PMID 14716844
- [Background] Vishnubhotla R, Sun S, Huq J, Bulic M, Ramesh A, Guzman G, Cho M, Glover SC. ROCK-II mediates colon cancer invasion via regulation of MMP-2 and MMP-13 at the site of invadopodia as revealed by multiphoton imaging. Lab Invest. 2007 Nov;87(11):1149-58. doi: 10.1038/labinvest.3700674. Epub 2007 Sep 17. PMID 17876296
- [Background] Kamai T, Tsujii T, Arai K, Takagi K, Asami H, Ito Y, Oshima H. Significant association of Rho/ROCK pathway with invasion and metastasis of bladder cancer. Clin Cancer Res. 2003 Jul;9(7):2632-41. PMID 12855641
- [Background] Sahai E, Marshall CJ. ROCK and Dia have opposing effects on adherens junctions downstream of Rho. Nat Cell Biol. 2002 Jun;4(6):408-15. doi: 10.1038/ncb796. PMID 11992112
- [Background] Croft DR, Sahai E, Mavria G, Li S, Tsai J, Lee WM, Marshall CJ, Olson MF. Conditional ROCK activation in vivo induces tumor cell dissemination and angiogenesis. Cancer Res. 2004 Dec 15;64(24):8994-9001. doi: 10.1158/0008-5472.CAN-04-2052. PMID 15604264
- [Background] Mizukami Y, Fujiki K, Duerr EM, Gala M, Jo WS, Zhang X, Chung DC. Hypoxic regulation of vascular endothelial growth factor through the induction of phosphatidylinositol 3-kinase/Rho/ROCK and c-Myc. J Biol Chem. 2006 May 19;281(20):13957-63. doi: 10.1074/jbc.M511763200. Epub 2006 Mar 16. PMID 16543245
- [Background] Somlyo AV, Phelps C, Dipierro C, Eto M, Read P, Barrett M, Gibson JJ, Burnitz MC, Myers C, Somlyo AP. Rho kinase and matrix metalloproteinase inhibitors cooperate to inhibit angiogenesis and growth of human prostate cancer xenotransplants. FASEB J. 2003 Feb;17(2):223-34. doi: 10.1096/fj.02-0655com. PMID 12554701
- [Background] Somlyo AV, Bradshaw D, Ramos S, Murphy C, Myers CE, Somlyo AP. Rho-kinase inhibitor retards migration and in vivo dissemination of human prostate cancer cells. Biochem Biophys Res Commun. 2000 Mar 24;269(3):652-9. doi: 10.1006/bbrc.2000.2343. PMID 10720471
- [Background] Ying H, Biroc SL, Li WW, Alicke B, Xuan JA, Pagila R, Ohashi Y, Okada T, Kamata Y, Dinter H. The Rho kinase inhibitor fasudil inhibits tumor progression in human and rat tumor models. Mol Cancer Ther. 2006 Sep;5(9):2158-64. doi: 10.1158/1535-7163.MCT-05-0440. PMID 16985048
- [Background] Bourguignon LY, Zhu H, Shao L, Zhu D, Chen YW. Rho-kinase (ROK) promotes CD44v(3,8-10)-ankyrin interaction and tumor cell migration in metastatic breast cancer cells. Cell Motil Cytoskeleton. 1999;43(4):269-87. doi: 10.1002/(SICI)1097-0169(1999)43:43.0.CO;2-5. PMID 10423269
- [Background] Barreiro O, Yanez-Mo M, Serrador JM, Montoya MC, Vicente-Manzanares M, Tejedor R, Furthmayr H, Sanchez-Madrid F. Dynamic interaction of VCAM-1 and ICAM-1 with moesin and ezrin in a novel endothelial docking structure for adherent leukocytes. J Cell Biol. 2002 Jun 24;157(7):1233-45. doi: 10.1083/jcb.200112126. Epub 2002 Jun 24. PMID 12082081
- [Background] Bivalacqua TJ, Champion HC, Usta MF, Cellek S, Chitaley K, Webb RC, Lewis RL, Mills TM, Hellstrom WJ, Kadowitz PJ. RhoA/Rho-kinase suppresses endothelial nitric oxide synthase in the penis: a mechanism for diabetes-associated erectile dysfunction. Proc Natl Acad Sci U S A. 2004 Jun 15;101(24):9121-6. doi: 10.1073/pnas.0400520101. Epub 2004 Jun 7. PMID 15184671
- [Background] Ming XF, Viswambharan H, Barandier C, Ruffieux J, Kaibuchi K, Rusconi S, Yang Z. Rho GTPase/Rho kinase negatively regulates endothelial nitric oxide synthase phosphorylation through the inhibition of protein kinase B/Akt in human endothelial cells. Mol Cell Biol. 2002 Dec;22(24):8467-77. doi: 10.1128/MCB.22.24.8467-8477.2002. PMID 12446767
- [Background] Tominaga T, Sugie K, Hirata M, Morii N, Fukata J, Uchida A, Imura H, Narumiya S. Inhibition of PMA-induced, LFA-1-dependent lymphocyte aggregation by ADP ribosylation of the small molecular weight GTP binding protein, rho. J Cell Biol. 1993 Mar;120(6):1529-37. doi: 10.1083/jcb.120.6.1529. PMID 7680658
- [Background] Sanchez-Madrid F, del Pozo MA. Leukocyte polarization in cell migration and immune interactions. EMBO J. 1999 Feb 1;18(3):501-11. doi: 10.1093/emboj/18.3.501. PMID 9927410
- [Background] Alevriadou BR. CAMs and Rho small GTPases: gatekeepers for leukocyte transendothelial migration. Focus on "VCAM-1-mediated Rac signaling controls endothelial cell-cell contacts and leukocyte transmigration". Am J Physiol Cell Physiol. 2003 Aug;285(2):C250-2. doi: 10.1152/ajpcell.00189.2003. No abstract available. PMID 12842833
- [Background] Etienne S, Adamson P, Greenwood J, Strosberg AD, Cazaubon S, Couraud PO. ICAM-1 signaling pathways associated with Rho activation in microvascular brain endothelial cells. J Immunol. 1998 Nov 15;161(10):5755-61. PMID 9820557
- [Background] Zhu F, Zhang Z, Wu G, Li Z, Zhang R, Ren J, Nong L. Rho kinase inhibitor fasudil suppresses migration and invasion though down-regulating the expression of VEGF in lung cancer cell line A549. Med Oncol. 2011 Jun;28(2):565-71. doi: 10.1007/s12032-010-9468-5. Epub 2010 Mar 19. PMID 20300976
- [Background] Nakabayashi H, Shimizu K. HA1077, a Rho kinase inhibitor, suppresses glioma-induced angiogenesis by targeting the Rho-ROCK and the mitogen-activated protein kinase kinase/extracellular signal-regulated kinase (MEK/ERK) signal pathways. Cancer Sci. 2011 Feb;102(2):393-9. doi: 10.1111/j.1349-7006.2010.01794.x. Epub 2010 Dec 19. PMID 21166955
- [Background] Washida N, Wakino S, Tonozuka Y, Homma K, Tokuyama H, Hara Y, Hasegawa K, Minakuchi H, Fujimura K, Hosoya K, Hayashi K, Itoh H. Rho-kinase inhibition ameliorates peritoneal fibrosis and angiogenesis in a rat model of peritoneal sclerosis. Nephrol Dial Transplant. 2011 Sep;26(9):2770-9. doi: 10.1093/ndt/gfr012. Epub 2011 Mar 4. PMID 21378147
- [Background] Kuno M, Takai S, Matsushima-Nishiwaki R, Minamitani C, Mizutani J, Otsuka T, Harada A, Adachi S, Kozawa O, Tokuda H. Rho-kinase inhibitors decrease TGF-beta-stimulated VEGF synthesis through stress-activated protein kinase/c-Jun N-terminal kinase in osteoblasts. Biochem Pharmacol. 2009 Jan 15;77(2):196-203. doi: 10.1016/j.bcp.2008.10.014. Epub 2008 Oct 19. PMID 18996357
- [Background] Takata K, Morishige K, Takahashi T, Hashimoto K, Tsutsumi S, Yin L, Ohta T, Kawagoe J, Takahashi K, Kurachi H. Fasudil-induced hypoxia-inducible factor-1alpha degradation disrupts a hypoxia-driven vascular endothelial growth factor autocrine mechanism in endothelial cells. Mol Cancer Ther. 2008 Jun;7(6):1551-61. doi: 10.1158/1535-7163.MCT-07-0428. PMID 18566226
- [Background] Hata Y, Miura M, Nakao S, Kawahara S, Kita T, Ishibashi T. Antiangiogenic properties of fasudil, a potent Rho-Kinase inhibitor. Jpn J Ophthalmol. 2008 Jan-Feb;52(1):16-23. doi: 10.1007/s10384-007-0487-5. Epub 2008 Mar 28. PMID 18369695
- [Background] Liu C, Li Y, Yu J, Feng L, Hou S, Liu Y, Guo M, Xie Y, Meng J, Zhang H, Xiao B, Ma C. Targeting the shift from M1 to M2 macrophages in experimental autoimmune encephalomyelitis mice treated with fasudil. PLoS One. 2013;8(2):e54841. doi: 10.1371/journal.pone.0054841. Epub 2013 Feb 13. PMID 23418431
- [Background] Ozeki K, Tanida S, Morimoto C, Inoue Y, Mizoshita T, Tsukamoto H, Shimura T, Kataoka H, Kamiya T, Nishiwaki E, Ishiguro H, Higashiyama S, Joh T. Telmisartan inhibits cell proliferation by blocking nuclear translocation of ProHB-EGF C-terminal fragment in colon cancer cells. PLoS One. 2013;8(2):e56770. doi: 10.1371/journal.pone.0056770. Epub 2013 Feb 22. PMID 23451083
- [Background] Sharpe M, Jarvis B, Goa KL. Telmisartan: a review of its use in hypertension. Drugs. 2001;61(10):1501-29. doi: 10.2165/00003495-200161100-00009. PMID 11558835
- [Background] Smith DH, Matzek KM, Kempthorne-Rawson J. Dose response and safety of telmisartan in patients with mild to moderate hypertension. J Clin Pharmacol. 2000 Dec;40(12 Pt 1):1380-90. PMID 11185637
- [Background] Stangier J, Su CA, Roth W. Pharmacokinetics of orally and intravenously administered telmisartan in healthy young and elderly volunteers and in hypertensive patients. J Int Med Res. 2000 Jul-Aug;28(4):149-67. doi: 10.1177/147323000002800401. PMID 11014323
- [Background] Forclaz A, Maillard M, Nussberger J, Brunner HR, Burnier M. Angiotensin II receptor blockade: is there truly a benefit of adding an ACE inhibitor? Hypertension. 2003 Jan;41(1):31-6. doi: 10.1161/01.hyp.0000047512.58862.a9. PMID 12511526
- [Background] Levine JE, Paczesny S, Sarantopoulos S. Clinical applications for biomarkers of acute and chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2012 Jan;18(1 Suppl):S116-24. doi: 10.1016/j.bbmt.2011.10.019. PMID 22226094
- [Background] Paczesny S. Discovery and validation of graft-versus-host disease biomarkers. Blood. 2013 Jan 24;121(4):585-94. doi: 10.1182/blood-2012-08-355990. Epub 2012 Nov 19. PMID 23165480
- [Background] Levine JE, Logan BR, Wu J, Alousi AM, Bolanos-Meade J, Ferrara JL, Ho VT, Weisdorf DJ, Paczesny S. Acute graft-versus-host disease biomarkers measured during therapy can predict treatment outcomes: a Blood and Marrow Transplant Clinical Trials Network study. Blood. 2012 Apr 19;119(16):3854-60. doi: 10.1182/blood-2012-01-403063. Epub 2012 Mar 1. PMID 22383800
- [Background] Vander Lugt MT, Braun TM, Hanash S, Ritz J, Ho VT, Antin JH, Zhang Q, Wong CH, Wang H, Chin A, Gomez A, Harris AC, Levine JE, Choi SW, Couriel D, Reddy P, Ferrara JL, Paczesny S. ST2 as a marker for risk of therapy-resistant graft-versus-host disease and death. N Engl J Med. 2013 Aug 8;369(6):529-39. doi: 10.1056/NEJMoa1213299. PMID 23924003
- [Background] Mueller T, Dieplinger B. The Presage((R)) ST2 Assay: analytical considerations and clinical applications for a high-sensitivity assay for measurement of soluble ST2. Expert Rev Mol Diagn. 2013 Jan;13(1):13-30. doi: 10.1586/erm.12.128. PMID 23256700
- [Background] Ferrara JL, Harris AC, Greenson JK, Braun TM, Holler E, Teshima T, Levine JE, Choi SW, Huber E, Landfried K, Akashi K, Vander Lugt M, Reddy P, Chin A, Zhang Q, Hanash S, Paczesny S. Regenerating islet-derived 3-alpha is a biomarker of gastrointestinal graft-versus-host disease. Blood. 2011 Dec 15;118(25):6702-8. doi: 10.1182/blood-2011-08-375006. Epub 2011 Oct 6. PMID 21979939
- [Background] Holler E, Landfried K, Meier J, Hausmann M, Rogler G. The role of bacteria and pattern recognition receptors in GVHD. Int J Inflam. 2010 Oct 31;2010:814326. doi: 10.4061/2010/814326. PMID 21188220
- [Background] Penack O, Holler E, van den Brink MR. Graft-versus-host disease: regulation by microbe-associated molecules and innate immune receptors. Blood. 2010 Mar 11;115(10):1865-72. doi: 10.1182/blood-2009-09-242784. Epub 2009 Dec 30. PMID 20042727
- [Background] Cooke KR, Gerbitz A, Crawford JM, Teshima T, Hill GR, Tesolin A, Rossignol DP, Ferrara JL. LPS antagonism reduces graft-versus-host disease and preserves graft-versus-leukemia activity after experimental bone marrow transplantation. J Clin Invest. 2001 Jun;107(12):1581-9. doi: 10.1172/JCI12156. PMID 11413166
- [Background] Lv M, Ye HG, Zhao XS, Zhao XY, Chang YJ, Liu DH, Xu LP, Huang XJ. Ceruloplasmin is a potential biomarker for aGvHD following allogeneic hematopoietic stem cell transplantation. PLoS One. 2013;8(3):e58735. doi: 10.1371/journal.pone.0058735. Epub 2013 Mar 7. PMID 23505556
- [Background] Romaschin AD, Klein DJ, Marshall JC. Bench-to-bedside review: Clinical experience with the endotoxin activity assay. Crit Care. 2012 Dec 3;16(6):248. doi: 10.1186/cc11495. PMID 23206992
- [Background] Hilmi I, Kellum J, Planinsic R, Foster D, Abdullah A, Damian D, Gligor S, Klein D, Abu-elmagd K. Endotoxemia is common following abdominal organ transplantation and is associated with reperfusion and rejection.Journal of Organ Dysfunction. Dec 2009, Vol. 5 Issue 4, p254-260.
- [Background] Sanada Y, Mizuta K, Urahashi T, Ihara Y, Wakiya T, Okada N, Yamada N, Ushijima K, Otomo S, Sakamoto K, Yasuda Y, Kawarasaki H. Impact of endotoxin measured by an endotoxin activity assay during liver transplantation. J Surg Res. 2013 Apr;180(2):349-55. doi: 10.1016/j.jss.2012.05.004. Epub 2012 May 24. PMID 22677614
- [Background] Marshall JC, Foster D, Vincent JL, Cook DJ, Cohen J, Dellinger RP, Opal S, Abraham E, Brett SJ, Smith T, Mehta S, Derzko A, Romaschin A; MEDIC study. Diagnostic and prognostic implications of endotoxemia in critical illness: results of the MEDIC study. J Infect Dis. 2004 Aug 1;190(3):527-34. doi: 10.1086/422254. Epub 2004 Jul 2. PMID 15243928
- [Background] Ikeda T, Ikeda K, Suda S, Ueno T. Usefulness of the endotoxin activity assay as a biomarker to assess the severity of endotoxemia in critically ill patients. Innate Immun. 2014 Nov;20(8):881-7. doi: 10.1177/1753425913516885. Epub 2014 Jan 7. PMID 24398861
- [Background] Jenq RR, Ubeda C, Taur Y, Menezes CC, Khanin R, Dudakov JA, Liu C, West ML, Singer NV, Equinda MJ, Gobourne A, Lipuma L, Young LF, Smith OM, Ghosh A, Hanash AM, Goldberg JD, Aoyama K, Blazar BR, Pamer EG, van den Brink MR. Regulation of intestinal inflammation by microbiota following allogeneic bone marrow transplantation. J Exp Med. 2012 May 7;209(5):903-11. doi: 10.1084/jem.20112408. Epub 2012 Apr 30. PMID 22547653
- [Background] Fricke WF, Maddox C, Song Y, Bromberg JS. Human microbiota characterization in the course of renal transplantation. Am J Transplant. 2014 Feb;14(2):416-27. doi: 10.1111/ajt.12588. Epub 2013 Dec 26. PMID 24373208
- [Background] Arck P, Handjiski B, Hagen E, Pincus M, Bruenahl C, Bienenstock J, Paus R. Is there a 'gut-brain-skin axis'? Exp Dermatol. 2010 May;19(5):401-5. doi: 10.1111/j.1600-0625.2009.01060.x. Epub 2010 Jan 25. PMID 20113345
- [Background] Gomez A, Hammer S, Braun T, Hanash S, Ferrara J, Greenson J, Wang H, Zhang Q, Vander Lugt M, Pongtornpipat P, Lamiman K, Colon M, Chang L, Choi S, Levine J, Harris A, Couriel D, Reddy P, Paczesny S. A novel CD4+CD146+CCR5+ T-cell population is a biomarker of intestinal graft-versus-host disease. 39th meeting of the European Group for Blood and Marrow Transplantation Wednesday, April 10, 2013, 09:30 - 09:42
- [Background] Cheng CI, Lin YC, Tsai TH, Lin HS, Liou CW, Chang WN, Lu CH, Yuen CM, Yip HK. The prognostic values of leukocyte Rho kinase activity in acute ischemic stroke. Biomed Res Int. 2014;2014:214587. doi: 10.1155/2014/214587. Epub 2014 Feb 27. PMID 24716192
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Patel PA, Patravale VB, Commercial Telmisartan Tablets: A Comparative Evaluation with Innovator Brand Micardis, International Journal of Pharma Sciences and Research (IJPSR) 2010, 1(8): 282-292.
- [Background] Michel MC, Bohner H, Koster J, Schafers R, Heemann U. Safety of telmisartan in patients with arterial hypertension : an open-label observational study. Drug Saf. 2004;27(5):335-44. doi: 10.2165/00002018-200427050-00005. PMID 15061687
- [Background] Schumacher H, Mancia G. The safety profile of telmisartan as monotherapy or combined with hydrochlorothiazide: a retrospective analysis of 50 studies. Blood Press Suppl. 2008 Jun;1:32-40. doi: 10.1080/08038020802144383. PMID 18705533
- [Background] Bahr IN, Tretter P, Kruger J, Stark RG, Schimkus J, Unger T, Kappert K, Scholze J, Parhofer KG, Kintscher U. High-dose treatment with telmisartan induces monocytic peroxisome proliferator-activated receptor-gamma target genes in patients with the metabolic syndrome. Hypertension. 2011 Oct;58(4):725-32. doi: 10.1161/HYPERTENSIONAHA.111.173542. Epub 2011 Aug 29. PMID 21876071
- [Background] Chetty VT, Damjanovic S, Gerstein H, Singh N, Yusuf S, Anand SS, Sharma AM. Metabolic effects of telmisartan in subjects with abdominal obesity: a prospective randomized controlled trial. Blood Press. 2014 Feb;23(1):54-60. doi: 10.3109/08037051.2013.791411. Epub 2013 Jun 3. PMID 23731019
- [Background] White WB. Comparative effects of telmisartan in the treatment of hypertension. J Clin Hypertens (Greenwich). 2002 Jul-Aug;4(4 Suppl 1):20-5. doi: 10.1111/j.1524-6175.2002.01585.x. PMID 12147925

RESULTS

PARTICIPANT FLOW:
Groups:
- 160 mg Telmisartan: 60 patients will receive 160 of Telmisartan (2 80 mg tablets) for 101 days
  Telmisartan
Period: Overall Study
Arm/Group | 160 mg Telmisartan
Started | 32
Completed | 21
Not Completed | 11
Not completed — Screen Failure | 3
Not completed — Withdrawal by Subject | 6
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Patients receiving Investigational Product not including screen failures
Arm/Group | 160 mg Telmisartan
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: Years] | 54.33 [23.51 to 73.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 or Greater Acute Graft vs. Host Disease (GVHD) in Patients Receiving Allogeneic HCT.
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | 160 mg Telmisartan
Number analyzed (Participants) | 27
Participants | 1

2. Secondary Outcome: Number of Subjects With Grade III-IV Hypotension as Per the National Cancer Institute's Common Terminology
Time Frame: 180 days post- transplant
Measure: Count of Participants; unit: Participants
Arm/Group | 160 mg Telmisartan
Number analyzed (Participants) | 27
Participants | 6

ADVERSE EVENTS:
Time Frame: From time of consent through +180 days post transplant
Arm/Group | 160 mg Telmisartan
All-Cause Mortality (participants affected / at risk) | 6/29
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 24/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 160 mg Telmisartan (N=29)
Pain (General disorders) | 1 (1)
Hospitalization (General disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Primary Graft Failure (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 160 mg Telmisartan (N=29)
Abdominal Cramping (Gastrointestinal disorders) | 2 (2)
Abdominal Pail (Gastrointestinal disorders) | 2 (2)
Acute GVHD (Immune system disorders) | 1 (1)
Acute GVHD (GI) (Immune system disorders) | 1 (1)
Acute GVHD (Liver) (Immune system disorders) | 1 (1)
Acute GVHD (Skin and GI) (Immune system disorders) | 1 (1)
Acute GVHD (Skin) (Immune system disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Acute Mental Status Change (Nervous system disorders) | 1 (1)
Adeno Viremia (Infections and infestations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1)
BK Viremia (Infections and infestations) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Chronic GVHD (Immune system disorders) | 2 (2)
Chronic GVHD (skin/liver, ocular, oral mucosa) (Immune system disorders) | 1 (1)
CMV Reactivation (Infections and infestations) | 1 (1)
CMV Viremia (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 3 (4)
Cystitis (Renal and urinary disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Delayed Engraftment (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Diarrhea (Intermittent) (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dizziness (Intermittent) (Nervous system disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea on Exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Early Satiety (Metabolism and nutrition disorders) | 1 (1)
Edema BLE (General disorders) | 1 (1)
Epstein-Barr Virus (Infections and infestations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
GVHD (GI) (Immune system disorders) | 3 (3)
GVHD (Liver) (Immune system disorders) | 2 (2)
GVHD (Oral) (Immune system disorders) | 1 (2)
GVHD (Skin) (Immune system disorders) | 5 (6)
GVHD (Skin/Liver) (Immune system disorders) | 1 (1)
H Pylori (Infections and infestations) | 1 (1)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Intermittent) (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypertension (Intermittent) (Vascular disorders) | 1 (1)
Hypoglycemia (intermittent) (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 12 (16)
Infection (Kidney) (Infections and infestations) | 1 (1)
Infection/Infestation (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (7)
Nausea (Intermittent) (Gastrointestinal disorders) | 2 (2)
Neutrophil Count Decreased (Investigations) | 1 (2)
Nocturia (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Erythematous) (Skin and subcutaneous tissue disorders) | 1 (2)
Rash on Upper Back (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory infection (HAP) (Infections and infestations) | 1 (1)
Right lower quadrant pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacral Decub (Skin and subcutaneous tissue disorders) | 1 (1)
Streptococcus mitis (Infections and infestations) | 3 (3)
Swelling R knee (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Vaginal abscess (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT02338232/Prot_SAP_000.pdf